CLINICAL TRIAL: NCT06572982
Title: Extension Study, Pilot, Single-arm, Compassionate Use of Hikma Azacitidine 300 mg Film Coated Tablets Test Product for the Acute Myeloid Leukaemia (AML) Patients Who Completed Hikma Bioequivalence Study With Protocol Number: HIK-AZA-2023-01
Brief Title: Extension Study, Pilot, Compassionate Use of Azacitidine 300 mg Film Coated Tablets for Acute Myeloid Leukaemia (AML) Patients
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hikma Pharmaceuticals LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HIK-AZA-2024-01
Record Dates: First submitted 2024-08-22; First posted 2024-08-27 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2025-09

CONDITIONS: Acute Myeloid Leukemia
Keywords: oral azacitidine; azacitidine; Acute Myeloid Leukaemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Azacitidine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Azacitidine 300 mg Film coated tablets (Experimental): Azacitidine 300 mg Film coated tablets
  Interventions: Drug: Azacitidine

INTERVENTIONS:
Drug: Azacitidine — 300 mg Film coated tablets

SUMMARY:
Extension study, pilot, single-arm, compassionate use of Hikma Azacitidine 300 mg Film coated tablets test product for the Acute Myeloid Leukaemia (AML) patients who completed Hikma bioequivalence study with protocol number: HIK-AZA-2023-01

ELIGIBILITY:
Inclusion Criteria:

1. Patients with AML who completed Hikma bioequivalence study of the same Hikma generic oral Azacitidine test product with protocol number: HIK-AZA-2023-01, and who consent to participate in the study.
2. Patients who understand and voluntarily sign a written informed consent document prior to any study related assessment/procedures are conducted.

Exclusion Criteria:

1. Female patients who are pregnant or nursing (lactating).
2. Patients with medical condition, laboratory abnormality, or psychiatric illness that, in the opinion of the investigator, might interfere with subject safety, compliance or evaluation of the condition of the study.
3. Patients with experience in any investigational drug in a clinical study within 6 months prior to study (except for patients who were enrolled in the Hikma Azacitidine bioequivalence study with protocol number: HIK-AZA-2023-01).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-04-29 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Descriptive statistics for the type, frequency, severity, expectedness, seriousness, outcome and relationship of adverse events to study drug | Up to 12 months
  Descriptive statistics for the type, frequency, severity, expectedness, seriousness, outcome and relationship of adverse events to study drug

CONTACTS AND LOCATIONS:
Locations (1):
- Sheikh Shakhbout Medical City, Abu Dhabi, United Arab Emirates

IPD SHARING:
Plan to Share IPD: No